CLINICAL TRIAL: NCT00603980
Title: Abuse Liability Study of Staccato® Alprazolam for Inhalation in Subjects With Histories of Sedative Abuse
Brief Title: Staccato Alprazolam Abuse Liability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-002-102; 22 January 2008
Record Dates: First submitted 2008-01-17; First posted 2008-01-29 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2009-01

CONDITIONS: Abuse Liability of Staccato Alprazolam
MeSH Terms: interventions — Alprazolam

STUDY DESIGN:
Intervention Model Description: The crossover schedule is planned according to a 7-treatment, 7-period Latin Square design due to E.J. Williams (1949), which is balanced for first-order carryover effects (Fleiss, 1986). Each subject will receive all treatments in this 7-treatment, 7- period Williams Square crossover design as suggested by Chen & Tsong (2007). This Williams Square will include one replication by 1 subject of each of the 14 sequences
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In order to reduce discrimination between placebo and active Staccato Alprazolam, taste blinding will be accomplished using a rapidly dissolving, intensely flavored product (candy, strip or breath spray). The product will be administered immediately after each oral capsule dosing (at the -60-min and 0- min time points).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Treatment sequence 1 (Other): Sequence 1: Q, 1, 2, 7, 3, 6, 4, 5; where Q=Qualifying sessions (2 mg oral alprazolam and placebo in random order), 1=placebo, 2=oral alprazolam 1 mg, 3= oral alprazolam 2 mg, 4= oral alprazolam 4 mg, 5= inhaled alprazolam 0.5 mg, 6= inhaled alprazolam 1 mg, 7= inhaled alprazolam 2 mg
  Interventions: Drug: Inhaled placebo + oral placebo; Drug: Inhaled alprazolam 0.5 mg; Drug: Inhaled alprazolam 1 mg; Drug: Inhaled alprazolam 2 mg; Drug: Oral alprazolam 1 mg; Drug: Oral alprazolam 2 mg; Drug: Oral alprazolam 4 m; Drug: Oral alprazolam 2 mg qualifying session; Drug: Oral placebo qualifying session
- Treatment sequence 2 (Other): Sequence Q, 2: 2, 3, 1, 4, 7, 5, 6; where Q=Qualifying sessions (2 mg oral alprazolam and placebo in random order), 1=placebo, 2=oral alprazolam 1 mg, 3= oral alprazolam 2 mg, 4= oral alprazolam 4 mg, 5= inhaled alprazolam 0.5 mg, 6= inhaled alprazolam 1 mg, 7= inhaled alprazolam 2 mg
  Interventions: Drug: Inhaled placebo + oral placebo; Drug: Inhaled alprazolam 0.5 mg; Drug: Inhaled alprazolam 1 mg; Drug: Inhaled alprazolam 2 mg; Drug: Oral alprazolam 1 mg; Drug: Oral alprazolam 2 mg; Drug: Oral alprazolam 4 m; Drug: Oral alprazolam 2 mg qualifying session; Drug: Oral placebo qualifying session
- Treatment sequence 3 (Other): Sequence 3: Q, 3, 4, 2, 5, 1, 6, 7; where Q=Qualifying sessions (2 mg oral alprazolam and placebo in random order), 1=placebo, 2=oral alprazolam 1 mg, 3= oral alprazolam 2 mg, 4= oral alprazolam 4 mg, 5= inhaled alprazolam 0.5 mg, 6= inhaled alprazolam 1 mg, 7= inhaled alprazolam 2 mg
  Interventions: Drug: Inhaled placebo + oral placebo; Drug: Inhaled alprazolam 0.5 mg; Drug: Inhaled alprazolam 1 mg; Drug: Inhaled alprazolam 2 mg; Drug: Oral alprazolam 1 mg; Drug: Oral alprazolam 2 mg; Drug: Oral alprazolam 4 m; Drug: Oral alprazolam 2 mg qualifying session; Drug: Oral placebo qualifying session
- Treatment sequence 4 (Other): Sequence 4: Q, 4, 5, 3, 6, 2, 7, 1; where Q=Qualifying sessions (2 mg oral alprazolam and placebo in random order), 1=placebo, 2=oral alprazolam 1 mg, 3= oral alprazolam 2 mg, 4= oral alprazolam 4 mg, 5= inhaled alprazolam 0.5 mg, 6= inhaled alprazolam 1 mg, 7= inhaled alprazolam 2 mg
  Interventions: Drug: Inhaled placebo + oral placebo; Drug: Inhaled alprazolam 0.5 mg; Drug: Inhaled alprazolam 1 mg; Drug: Inhaled alprazolam 2 mg; Drug: Oral alprazolam 1 mg; Drug: Oral alprazolam 2 mg; Drug: Oral alprazolam 4 m; Drug: Oral alprazolam 2 mg qualifying session; Drug: Oral placebo qualifying session
- Treatment sequence 5 (Other): Sequence 5: Q, 5, 6, 4, 7, 3, 1, 2; where Q=Qualifying sessions (2 mg oral alprazolam and placebo in random order), 1=placebo, 2=oral alprazolam 1 mg, 3= oral alprazolam 2 mg, 4= oral alprazolam 4 mg, 5= inhaled alprazolam 0.5 mg, 6= inhaled alprazolam 1 mg, 7= inhaled alprazolam 2 mg
  Interventions: Drug: Inhaled placebo + oral placebo; Drug: Inhaled alprazolam 0.5 mg; Drug: Inhaled alprazolam 1 mg; Drug: Inhaled alprazolam 2 mg; Drug: Oral alprazolam 1 mg; Drug: Oral alprazolam 2 mg; Drug: Oral alprazolam 4 m; Drug: Oral alprazolam 2 mg qualifying session; Drug: Oral placebo qualifying session
- Treatment sequence 6 (Other): Sequence 6: Q, 6, 7, 5, 1, 4, 2, 3; where Q=Qualifying sessions (2 mg oral alprazolam and placebo in random order), 1=placebo, 2=oral alprazolam 1 mg, 3= oral alprazolam 2 mg, 4= oral alprazolam 4 mg, 5= inhaled alprazolam 0.5 mg, 6= inhaled alprazolam 1 mg, 7= inhaled alprazolam 2 mg
  Interventions: Drug: Inhaled placebo + oral placebo; Drug: Inhaled alprazolam 0.5 mg; Drug: Inhaled alprazolam 1 mg; Drug: Inhaled alprazolam 2 mg; Drug: Oral alprazolam 1 mg; Drug: Oral alprazolam 2 mg; Drug: Oral alprazolam 4 m; Drug: Oral alprazolam 2 mg qualifying session; Drug: Oral placebo qualifying session
- Treatment sequence 7 (Other): Sequence 7: Q, 7, 1, 6, 2, 5, 3, 4; where Q=Qualifying sessions (2 mg oral alprazolam and placebo in random order), 1=placebo, 2=oral alprazolam 1 mg, 3= oral alprazolam 2 mg, 4= oral alprazolam 4 mg, 5= inhaled alprazolam 0.5 mg, 6= inhaled alprazolam 1 mg, 7= inhaled alprazolam 2 mg
  Interventions: Drug: Inhaled placebo + oral placebo; Drug: Inhaled alprazolam 0.5 mg; Drug: Inhaled alprazolam 1 mg; Drug: Inhaled alprazolam 2 mg; Drug: Oral alprazolam 1 mg; Drug: Oral alprazolam 2 mg; Drug: Oral alprazolam 4 m; Drug: Oral alprazolam 2 mg qualifying session; Drug: Oral placebo qualifying session
- Treatment sequence 8 (Other): Sequence 8: Q, 5, 4, 6, 3, 7, 2, 1; where Q=Qualifying sessions (2 mg oral alprazolam and placebo in random order), 1=placebo, 2=oral alprazolam 1 mg, 3= oral alprazolam 2 mg, 4= oral alprazolam 4 mg, 5= inhaled alprazolam 0.5 mg, 6= inhaled alprazolam 1 mg, 7= inhaled alprazolam 2 mg
  Interventions: Drug: Inhaled placebo + oral placebo; Drug: Inhaled alprazolam 0.5 mg; Drug: Inhaled alprazolam 1 mg; Drug: Inhaled alprazolam 2 mg; Drug: Oral alprazolam 1 mg; Drug: Oral alprazolam 2 mg; Drug: Oral alprazolam 4 m; Drug: Oral alprazolam 2 mg qualifying session; Drug: Oral placebo qualifying session
- Treatment sequence 9 (Other): Sequence 9: Q, 6, 5, 7, 4, 1, 3, 2; where Q=Qualifying sessions (2 mg oral alprazolam and placebo in random order), 1=placebo, 2=oral alprazolam 1 mg, 3= oral alprazolam 2 mg, 4= oral alprazolam 4 mg, 5= inhaled alprazolam 0.5 mg, 6= inhaled alprazolam 1 mg, 7= inhaled alprazolam 2 mg
  Interventions: Drug: Inhaled placebo + oral placebo; Drug: Inhaled alprazolam 0.5 mg; Drug: Inhaled alprazolam 1 mg; Drug: Inhaled alprazolam 2 mg; Drug: Oral alprazolam 1 mg; Drug: Oral alprazolam 2 mg; Drug: Oral alprazolam 4 m; Drug: Oral alprazolam 2 mg qualifying session; Drug: Oral placebo qualifying session
- Treatment sequence 10 (Other): Sequence 10: Q, 7, 6, 1, 5, 2, 4, 3; where Q=Qualifying sessions (2 mg oral alprazolam and placebo in random order), 1=placebo, 2=oral alprazolam 1 mg, 3= oral alprazolam 2 mg, 4= oral alprazolam 4 mg, 5= inhaled alprazolam 0.5 mg, 6= inhaled alprazolam 1 mg, 7= inhaled alprazolam 2 mg
  Interventions: Drug: Inhaled placebo + oral placebo; Drug: Inhaled alprazolam 0.5 mg; Drug: Inhaled alprazolam 1 mg; Drug: Inhaled alprazolam 2 mg; Drug: Oral alprazolam 1 mg; Drug: Oral alprazolam 2 mg; Drug: Oral alprazolam 4 m; Drug: Oral alprazolam 2 mg qualifying session; Drug: Oral placebo qualifying session
- Treatment sequence 11 (Other): Sequence 11: Q, 1, 7, 2, 6, 3, 5, 4; where Q=Qualifying sessions (2 mg oral alprazolam and placebo in random order), 1=placebo, 2=oral alprazolam 1 mg, 3= oral alprazolam 2 mg, 4= oral alprazolam 4 mg, 5= inhaled alprazolam 0.5 mg, 6= inhaled alprazolam 1 mg, 7= inhaled alprazolam 2 mg
  Interventions: Drug: Inhaled placebo + oral placebo; Drug: Inhaled alprazolam 0.5 mg; Drug: Inhaled alprazolam 1 mg; Drug: Inhaled alprazolam 2 mg; Drug: Oral alprazolam 1 mg; Drug: Oral alprazolam 2 mg; Drug: Oral alprazolam 4 m; Drug: Oral alprazolam 2 mg qualifying session; Drug: Oral placebo qualifying session
- Treatment sequence 12 (Other): Sequence 12: Q, 2, 1, 3, 7, 4, 6, 5; where Q=Qualifying sessions (2 mg oral alprazolam and placebo in random order), 11=placebo, 2=oral alprazolam 1 mg, 3= oral alprazolam 2 mg, 4= oral alprazolam 4 mg, 5= inhaled alprazolam 0.5 mg, 6= inhaled alprazolam 1 mg, 7= inhaled alprazolam 2 mg
  Interventions: Drug: Inhaled placebo + oral placebo; Drug: Inhaled alprazolam 0.5 mg; Drug: Inhaled alprazolam 1 mg; Drug: Inhaled alprazolam 2 mg; Drug: Oral alprazolam 1 mg; Drug: Oral alprazolam 2 mg; Drug: Oral alprazolam 4 m; Drug: Oral alprazolam 2 mg qualifying session; Drug: Oral placebo qualifying session
- Treatment sequence 13 (Other): Sequence 13: Q, 3, 2, 4, 1, 5, 7, 6; where Q=Qualifying sessions (2 mg oral alprazolam and placebo in random order), 1=placebo, 2=oral alprazolam 1 mg, 3= oral alprazolam 2 mg, 4= oral alprazolam 4 mg, 5= inhaled alprazolam 0.5 mg, 6= inhaled alprazolam 1 mg, 7= inhaled alprazolam 2 mg
  Interventions: Drug: Inhaled placebo + oral placebo; Drug: Inhaled alprazolam 0.5 mg; Drug: Inhaled alprazolam 1 mg; Drug: Inhaled alprazolam 2 mg; Drug: Oral alprazolam 1 mg; Drug: Oral alprazolam 2 mg; Drug: Oral alprazolam 4 m; Drug: Oral alprazolam 2 mg qualifying session; Drug: Oral placebo qualifying session
- Treatment sequence 14 (Other): Sequence 14: Q, 4, 3, 5, 2, 6, 1, 7; where Q=Qualifying sessions (2 mg oral alprazolam and placebo in random order), 11=placebo, 2=oral alprazolam 1 mg, 3= oral alprazolam 2 mg, 4= oral alprazolam 4 mg, 5= inhaled alprazolam 0.5 mg, 6= inhaled alprazolam 1 mg, 7= inhaled alprazolam 2 mg
  Interventions: Drug: Inhaled placebo + oral placebo; Drug: Inhaled alprazolam 0.5 mg; Drug: Inhaled alprazolam 1 mg; Drug: Inhaled alprazolam 2 mg; Drug: Oral alprazolam 1 mg; Drug: Oral alprazolam 2 mg; Drug: Oral alprazolam 4 m; Drug: Oral alprazolam 2 mg qualifying session; Drug: Oral placebo qualifying session

INTERVENTIONS:
Drug: Inhaled placebo + oral placebo — Inhaled Staccato placebo + oral placebo
Drug: Inhaled alprazolam 0.5 mg — Inhaled Staccato alprazolam 0.5 mg + oral placebo
Drug: Inhaled alprazolam 1 mg — Inhaled Staccato alprazolam 1 mg + oral placebo
Drug: Inhaled alprazolam 2 mg — Inhaled Staccato alprazolam 2 mg + oral placebo
Drug: Oral alprazolam 1 mg — Oral alprazolam 1 mg + Inhaled placebo
Drug: Oral alprazolam 2 mg — Oral alprazolam 2 mg + Inhaled placebo
Drug: Oral alprazolam 4 m — Oral alprazolam 4 mg + Inhaled placebo
Drug: Oral alprazolam 2 mg qualifying session — Qualifying session (2 mg oral alprazolam)
Drug: Oral placebo qualifying session — Qualifying control session (oral placebo)

SUMMARY:
Compare the abuse liabilities of Staccato Alprazolam, oral immediate-release alprazolam, and Staccato Placebo.

DETAILED DESCRIPTION:
The Phase 1 clinical study compared the abuse liabilities of Staccato Alprazolam, oral immediate-release alprazolam, and Staccato Placebo in 14 subjects with a history of sedative abuse. Subjects who met the inclusion/exclusion criteria received 2 mg of oral alprazolam and matching placebo over 2 sessions. Those who demonstrated greater liking for alprazolam versus placebo were eligible to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18 to 55 years, inclusive, who have a history of substance abuse or dependence on barbiturates and/or benzodiazepine receptor agonists for their intoxicating effects

Exclusion Criteria:

* Subjects with a significant current psychiatric illness or taking any psychotropic prescription medications for therapeutic uses.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roland R Griffiths, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

REFERENCES:
- [Result] Reissig CJ, Harrison JA, Carter LP, Griffiths RR. Inhaled vs. oral alprazolam: subjective, behavioral and cognitive effects, and modestly increased abuse potential. Psychopharmacology (Berl). 2015 Mar;232(5):871-83. doi: 10.1007/s00213-014-3721-0. Epub 2014 Sep 9. PMID 25199955

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each participants was to receive all 7 interventions in a randomized order in a crossover design
Groups:
- All Subjects Entering: All subjects entering the crossover qualification period
Period: Study Qualification
Arm/Group | All Subjects Entering
Started | 31
Completed | 15
Not Completed | 16
Not completed — Protocol Violation | 3
Not completed — Inconsistent data reporting | 13
Period: Main Study
Arm/Group | All Subjects Entering
Started | 15
Completed | 14
Not Completed | 1
Not completed — 14th subject completed trial | 1

BASELINE CHARACTERISTICS:
Groups:
- Qualifying Session (Includes Crossover Group): All subjects received Placebo and Oral alprazolam 2 mg in a randomized order to Qualify
  Each subject was to receive all 7 interventions (Placebo, Oral alprazolam 1, 2 & 3 mg, Inhaled alprazolam 0.5, 1, & 2 mg) in a randomized order in a crossover design
Arm/Group | Qualifying Session (Includes Crossover Group)
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.032 (38.032)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Response to EDQ Question Number 5, "Rate the Degree to Which You Would Like to Take the Drug Again"
Description: The End of Day Questionnaire (EDQ) is a 7-question computerized instrument in which subjects rate the overall effect of the drug they received that day. The primary outcome measure for this trial is the categorical response to question number 5, "Rate the degree to which you would like to take the drug again", with a numerical value assigned to each of the responses allowed: 0=Not at all, 1=A little, 2=Moderately, 3=Quite a bit, 4=Very much
Time Frame: End of day for each of the 7 crossover treatments
Population: Efficacy (crossover) Population, n=14. LSM & SEM are based on all 14 subjects completing all 7 treatments. PROC MIXED model used assigns the same SEM to all 7 treatments.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Inhaled Staccato Placebo +oral placebo
- Oral Alprazolam 4 mg: Oral alprazolam 4 mg + inhaled placebo
- Inhaled Alprazolam 2 mg: Inhaled Staccato alprazolam 0.5 mg + oral placebo placebo
Arm/Group | Placebo | Oral Alprazolam 1 mg | Oral Alprazolam 2 mg | Oral Alprazolam 4 mg | Inhaled Alprazolam 0.5 mg | Inhaled Alprazolam 1 mg | Inhaled Alprazolam 2 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14
units on a scale | 0 (0.349) | 1.714 (0.349) | 2.143 (0.349) | 2.286 (0.349) | 1.00 (0.349) | 1.714 (0.349) | 2.214 (0.349)

2. Secondary Outcome: EDQ Question Number 2 "Rate Your Overall Liking of the Drug Effect"
Description: The within patient rank (1-7) of End of Day question number 2 (of primary interest), "Rate your overall liking of the drug effect", response options range from -4 to +4:
  * 4=Dislike very much
  * 3=Dislike quite a bit
  * 2=Dislike somewhat
  * 1=Dislike, but not very much 0=NEUTRAL OR NO EFFECT
    * 1=Like, but not very much
    * 2=Like somewhat
    * 3=Like quite a bit
    * 4=Like very much Thus a higher rank means a stronger drug effect and a lower rank a lesser drug effect
Time Frame: End of day for each of the 7 crossover treatments
Population: Efficacy (crossover) Population, n=14
  LS Means via SAS PROC MIXED non-parametric model (ranks within subject), treatment and period as fixed effects, ddf=72
  LSM & SEM are based on the ranks of scores within each subject across all 14 subjects completing all 7 treatments.
  PROC MIXED model assigns the same SEM to all 7 treatments.
Measure: Least Squares Mean (Standard Error); unit: Rank across the 7 treatments
Arm/Group | Placebo | Oral Alprazolam 1 mg | Oral Alprazolam 2 mg | Oral Alprazolam 4 mg | Inhaled Alprazolam 0.5 mg | Inhaled Alprazolam 1 mg | Inhaled Alprazolam 2 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14
Rank across the 7 treatments | 1.679 (0.349) | 4.214 (0.349) | 4.429 (0.349) | 4.607 (0.349) | 2.571 (0.349) | 4.857 (0.349) | 5.643 (0.349)

3. Secondary Outcome: EDQ Question Number 6 " Estimate the Amount of Money You Think the Drug You Took Today Would be Worth on the Street".
Description: EDQ question number 6 (of primary interest)," Estimate the amount of money you think the drug you took today would be worth on the street".
Time Frame: End of day for each of the 7 crossover treatments
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Dollars ($)
Arm/Group | Placebo | Oral Alprazolam 1 mg | Oral Alprazolam 2 mg | Oral Alprazolam 4 mg | Inhaled Alprazolam 0.5 mg | Inhaled Alprazolam 1 mg | Inhaled Alprazolam 2 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14
Dollars ($) | 1.750 (0.402) | 3.571 (0.402) | 7.071 (0.402) | 8.714 (0.402) | 2.857 (0.402) | 4.286 (0.402) | 8.571 (0.402)

4. Secondary Outcome: EDQ Question Number 1, "Rate the Overall Strength of the Drug Effect"
Description: The within patient rank (1-7) of End of Day question number 1, "Rate the overall strength of the drug effect", response options range from 0-4:
  0=No drug effect at all
  1. Possible mild effect, but not sure
  2. Definite mild effect
  3. Moderate strong drug effect
  4. Very strong drug effect Thus a higher rank means a stronger drug effect and a lower rank a lesser drug effect
Time Frame: End of day for each of the 7 crossover treatments
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Rank across the 7 treatments
Arm/Group | Placebo | Oral Alprazolam 1 mg | Oral Alprazolam 2 mg | Oral Alprazolam 4 mg | Inhaled Alprazolam 0.5 mg | Inhaled Alprazolam 1 mg | Inhaled Alprazolam 2 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14
Rank across the 7 treatments | 1.429 (0.317) | 3.536 (0.317) | 4.821 (0.317) | 5.429 (0.317) | 2.893 (0.317) | 4.143 (0.317) | 5.750 (0.317)

5. Secondary Outcome: EDQ Question Number 7,"What Would You be Willing to Pay for Today's Drug?"
Description: EDQ question number 7," What would you be willing to pay for today's drug?"
Time Frame: End of day for each of the 7 crossover treatments
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Dollars ($)
Arm/Group | Placebo | Oral Alprazolam 1 mg | Oral Alprazolam 2 mg | Oral Alprazolam 4 mg | Inhaled Alprazolam 0.5 mg | Inhaled Alprazolam 1 mg | Inhaled Alprazolam 2 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14
Dollars ($) | 1.607 (0.387) | 3.821 (0.387) | 4.571 (0.387) | 5.179 (0.387) | 2.964 (0.387) | 4.107 (0.387) | 5.750 (0.387)

6. Secondary Outcome: Maximum of DEQ Question 1 "Rate the Strength of the Drug Effect" (at the 10 Time Points, Predose Through 9 Hours)
Description: The within patient rank (1-7) of Drug Effect Questionnaire question number 1: Rate the STRENGTH of the drug effect you are feeling RIGHT NOW; response options range for 0 to 4:
  "No drug effect at all"=0, "Possible mild effect, but not sure"=1, "Definite mild effect"=2, "Moderate strong drug effect"=3, "Very strong drug effect"=4 Maximum of the 10 time points (predose through 9 hours) Thus a higher rank means a stronger drug effect and a lower rank a lesser drug effect
Time Frame: DEQ was assessed at the 10 time points (predose through 9 hours)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Rank across the 7 treatments
Arm/Group | Placebo | Oral Alprazolam 1 mg | Oral Alprazolam 2 mg | Oral Alprazolam 4 mg | Inhaled Alprazolam 0.5 mg | Inhaled Alprazolam 1 mg | Inhaled Alprazolam 2 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14
Rank across the 7 treatments | 1.571 (0.340) | 3.143 (0.340) | 4.714 (0.340) | 5.536 (0.340) | 3.036 (0.340) | 4.250 (0.340) | 5.750 (0.340)

7. Secondary Outcome: Maximum of DEQ Question 2 "Rate Your Liking of the Drug Effect" at the 10 Time Points (Predose Through 9 Hours)
Description: The within patient rank (1-7) of maximum of the Rate your LIKING of the drug effect you are feeling RIGHT NOW; response options range from -4 to +4:
  "Dislike very much"=-4, "Dislike quite a bit"=-3, "Dislike somewhat"=-2, "Dislike, but not very much"=-1, "NEUTRAL OR NO EFFECT"=0, "Like, but not very much"=1, "Like somewhat"=2, "Like quite a bit"=3, "Like very much"=4 Thus a higher rank means a stronger drug effect and a lower rank a lesser drug effect
Time Frame: DEQ was assessed at the 10 time points (predose through 9 hours)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Rank across the 7 treatments
Arm/Group | Placebo | Oral Alprazolam 1 mg | Oral Alprazolam 2 mg | Oral Alprazolam 4 mg | Inhaled Alprazolam 0.5 mg | Inhaled Alprazolam 1 mg | Inhaled Alprazolam 2 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14
Rank across the 7 treatments | 1.607 (0.343) | 3.500 (0.343) | 4.536 (0.343) | 5.536 (0.343) | 2.893 (0.343) | 4.250 (0.343) | 5.679 (0.343)

8. Secondary Outcome: Observer Rated Questionnaire 1) Maximum of Sedation/Sleepiness
Description: The within patient rank (1-7) of Maximum of Observer Rated Questionnaire (ORQ): A trained and blinded staff member completed observer ratings as the subject completed the questionnaires and psychomotor assessment testing at each time point.
  The observer rated the subject on sedation/sleepiness, muscle relaxation, impaired posture, impaired speech, confusion/disorientation, stimulation/arousal and strength of drug effect on a five-point scale from 0 (indicating normal or no effect) to 4 (indicating extreme drug effect).
  Maximum of the 10 time points (predose through 9 hours) Thus a higher rank means a stronger drug effect and a lower rank a lesser drug effect
Time Frame: ORQ was assessed at the 10 time points (predose through 9 hours)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Rank across the 7 treatments
Arm/Group | Placebo | Oral Alprazolam 1 mg | Oral Alprazolam 2 mg | Oral Alprazolam 4 mg | Inhaled Alprazolam 0.5 mg | Inhaled Alprazolam 1 mg | Inhaled Alprazolam 2 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14
Rank across the 7 treatments | 2.250 (0.313) | 3.679 (0.313) | 4.607 (0.313) | 4.714 (0.313) | 3.929 (0.313) | 4.000 (0.313) | 4.821 (0.313)

9. Secondary Outcome: Observer Rated Questionnaire 2) Maximum of Muscle Relaxation Locomotor
Description: The within patient rank (1-7) of maximum of the observer rated the subject on muscle relaxation (locomotor) on a five-point scale from 0 (indicating normal or no effect) to 4 (indicating extreme drug effect).
  Maximum of the 10 time points (predose through 9 hours) Thus a higher rank means a stronger drug effect and a lower rank a lesser drug effect
Time Frame: ORQ was assessed at the 10 time points (predose through 9 hours)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Rank across the 7 treatments
Arm/Group | Placebo | Oral Alprazolam 1 mg | Oral Alprazolam 2 mg | Oral Alprazolam 4 mg | Inhaled Alprazolam 0.5 mg | Inhaled Alprazolam 1 mg | Inhaled Alprazolam 2 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14
Rank across the 7 treatments | 2.464 (0.287) | 2.964 (0.287) | 4.643 (0.287) | 6.357 (0.287) | 2.821 (0.287) | 3.571 (0.287) | 5.179 (0.287)

10. Secondary Outcome: Observer Rated Questionnaire 3) Maximum of Muscle Relaxation Non-locomotor
Description: The within patient rank (1-7) of maximum of the observer rated the subject on muscle relaxation (non-locomotor) on a five-point scale from 0 (indicating normal or no effect) to 4 (indicating extreme drug effect).
  Thus a higher rank means a stronger drug effect and a lower rank a lesser drug effect
Time Frame: ORQ was assessed at the 10 time points (predose through 9 hours)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Oral Alprazolam 1 mg | Oral Alprazolam 2 mg | Oral Alprazolam 4 mg | Inhaled Alprazolam 0.5 mg | Inhaled Alprazolam 1 mg | Inhaled Alprazolam 2 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14
units on a scale | 2.536 (0.282) | 3.036 (0.282) | 4.607 (0.282) | 6.393 (0.282) | 2.714 (0.282) | 3.786 (0.282) | 4.929 (0.282)

11. Secondary Outcome: Observer Rated Questionnaire 4) Maximum of Muscle Relaxation Posture
Description: The within patient rank (1-7) of maximum of the observer rated the subject on muscle relaxation (posture) on a five-point scale from 0 (indicating normal or no effect) to 4 (indicating extreme drug effect).
  Thus a higher rank means a stronger drug effect and a lower rank a lesser drug effect
Time Frame: ORQ was assessed at the 10 time points (predose through 9 hours)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Rank across the 7 treatments
Arm/Group | Placebo | Oral Alprazolam 1 mg | Oral Alprazolam 2 mg | Oral Alprazolam 4 mg | Inhaled Alprazolam 0.5 mg | Inhaled Alprazolam 1 mg | Inhaled Alprazolam 2 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14
Rank across the 7 treatments | 2.750 (0.337) | 2.893 (0.337) | 3.964 (0.337) | 6.250 (0.337) | 2.929 (0.337) | 2.929 (0.337) | 2.929 (0.337)

12. Secondary Outcome: Observer Rated Questionnaire 5) Maximum of Speech
Description: The within patient rank (1-7) of maximum of the observer rated the subject on speech on a five-point scale from 0 (indicating normal or no effect) to 4 (indicating extreme drug effect).
  Thus a higher rank means a stronger drug effect and a lower rank a lesser drug effect
Time Frame: ORQ was assessed at the 10 time points (predose through 9 hours)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Rank across the 7 treatments
Arm/Group | Placebo | Oral Alprazolam 1 mg | Oral Alprazolam 2 mg | Oral Alprazolam 4 mg | Inhaled Alprazolam 0.5 mg | Inhaled Alprazolam 1 mg | Inhaled Alprazolam 2 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14
Rank across the 7 treatments | 2.214 (0.284) | 2.893 (0.284) | 4.786 (0.284) | 6.393 (0.284) | 3.071 (0.284) | 3.071 (0.284) | 5.357 (0.284)

13. Secondary Outcome: Observer Rated Questionnaire 6) Maximum of Confusion/Disorientation
Description: The within patient rank (1-7) of maximum of the observer rated the subject on Confusion/Disorientation on a five-point scale from 0 (indicating normal or no effect) to 4 (indicating extreme drug effect).
  Thus a higher rank means a stronger drug effect and a lower rank a lesser drug effect
Time Frame: ORQ was assessed at the 10 time points (predose through 9 hours)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Rank across the 7 treatments
Arm/Group | Placebo | Oral Alprazolam 1 mg | Oral Alprazolam 2 mg | Oral Alprazolam 4 mg | Inhaled Alprazolam 0.5 mg | Inhaled Alprazolam 1 mg | Inhaled Alprazolam 2 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14
Rank across the 7 treatments | 1.929 (0.282) | 2.821 (0.282) | 4.893 (0.282) | 6.429 (0.282) | 3.393 (0.282) | 3.107 (0.282) | 5.429 (0.282)

14. Secondary Outcome: Observer Rated Questionnaire 7) Maximum of Stimulation/Arousal
Description: The within patient rank (1-7) of maximum of the observer rated the subject on Stimulation/Arousal on a five-point scale from 0 (indicating normal or no effect) to 4 (indicating extreme drug effect).
  Thus a higher rank means a stronger drug effect and a lower rank a lesser drug effect
Time Frame: ORQ was assessed at the 10 time points (predose through 9 hours)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Rank across the 7 treatments
Arm/Group | Placebo | Oral Alprazolam 1 mg | Oral Alprazolam 2 mg | Oral Alprazolam 4 mg | Inhaled Alprazolam 0.5 mg | Inhaled Alprazolam 1 mg | Inhaled Alprazolam 2 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14
Rank across the 7 treatments | 3.964 (0.087) | 3.964 (0.087) | 3.964 (0.087) | 3.964 (0.087) | 3.964 (0.087) | 3.964 (0.087) | 4,214 (0.087)

15. Secondary Outcome: Observer Rated Questionnaire 8) Maximum of Drug Strength
Description: The within patient rank (1-7) of maximum of the observer rated the subject on Drug Strength on a five-point scale from 0 (indicating normal or no effect) to 4 (indicating extreme drug effect).
  Thus a higher rank means a stronger drug effect and a lower rank a lesser drug effect
Time Frame: ORQ was assessed at the 10 time points (predose through 9 hours)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Rank across the 7 treatments
Arm/Group | Oral Alprazolam 1 mg | Placebo | Oral Alprazolam 2 mg | Oral Alprazolam 4 mg | Inhaled Alprazolam 0.5 mg | Inhaled Alprazolam 1 mg | Inhaled Alprazolam 2 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14
Rank across the 7 treatments | 2.786 (0.286) | 1.714 (0.286) | 4.571 (0.286) | 6.321 (0.286) | 3.000 (0.286) | 3.929 (0.286) | 5.679 (0.286)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were considered treatment related from the first exposure to study treatment until 30 days after the last treatment
Description: Adverse events (AEs) were assessed at 14 pre-specified time points for the 24-hour period after dosing, as well as whenever spontaneously reported by the subjects or study staff
Groups:
- Qualifying Session 2 mg Oral: Qualifying session, 2 mg oral alprazolam
- Qualifying Session Oral Placebo: Qualifying session, oral placebo (alprazolam 0 mg)
Arm/Group | Placebo | Oral Alprazolam 1 mg | Oral Alprazolam 2 mg | Oral Alprazolam 4 mg | Inhaled Alprazolam 0.5 mg | Inhaled Alprazolam 1 mg | Inhaled Alprazolam 2 mg | Qualifying Session 2 mg Oral | Qualifying Session Oral Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/14 | 0/15 | 0/14 | 0/15 | 0/15 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/14 | 0/15 | 0/14 | 0/15 | 0/15 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/14 | 1/15 | 0/14 | 0/15 | 0/15 | 0/28 | 1/28
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Oral Alprazolam 1 mg (N=15) | Oral Alprazolam 2 mg (N=14) | Oral Alprazolam 4 mg (N=15) | Inhaled Alprazolam 0.5 mg (N=14) | Inhaled Alprazolam 1 mg (N=15) | Inhaled Alprazolam 2 mg (N=15) | Qualifying Session 2 mg Oral (N=28) | Qualifying Session Oral Placebo (N=28)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
A limitation of the current study was the lack of assessment of drug plasma levels. The differences in abuse potential measures may be due to differences in absorption, peak drug plasma levels, or other PK parameters

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less